CLINICAL TRIAL: NCT01462799
Title: COR-PRIM: Problem-based Learning in Patient Education After an Event of Coronary Heart Disease. A Randomised Study in Primary Care of Long-term Effects on Self-care
Brief Title: COR-PRIM: Problem-based Learning (PBL) After Coronary Heart Disease (CHD) - Long-term Evaluation in Primary Care of Self-care
Acronym: CORPRIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Linkoeping University (Other Government)
Collaborators: Swedish Heart Lung Foundation (Other); Ostergotland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Anita Karner, University Lecturer, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: COR-PRIM-Dnr 2010/128-3
Record Dates: First submitted 2011-10-24; First posted 2011-10-31 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-10

CONDITIONS: Coronary Heart Disease
Keywords: PBL; patient education; coronary heart disease; empowerment; self-efficacy; self-care; Focus on to determine the long term effectiveness of PBL in patient education by comparison of standardized homesent information in patients with CHD.; Further focus is on patients' self-care goals, beliefs, self-efficacy and empowerment to make lifestyle changes.
MeSH Terms: conditions — Coronary Disease; Empowerment | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PBL- patient education (Experimental): Patients will be randomised to PBL in patient education (experiment group)
  Interventions: Behavioral: PBL in patient education; Behavioral: Mailed patient information
- Mailed patient information (Experimental): Patients will be randomised to controlgroup receiving mailed patient information during the year
  Interventions: Behavioral: Mailed patient information

INTERVENTIONS:
Behavioral: PBL in patient education — The experiment group will enter a PBL patient education that is characterised by autonomous learning. The patients work together in small groups. Focus is on lifestyle changes. Starting point of learning is the patient's individual life style goals. Thirteen meetings during 1 year for 2 hours; weekly for the first month, every second week next two months and the last meetings 16, 20 and 26, 39 and 52 weeks after start. The programme shall be completed 1 year after start. The patients work with starting triggers such as pictures, texts, or concrete materials. Nurses work as tutors (after completion of a tutorial education) during the meetings using a problem based model to support patients formulate issues and goals to work with during the year. When the patients do not solve question the possibility of inviting e.g. a GP, dietician, pharmacist or physiotherapist is possible.
  Arms: PBL- patient education
Behavioral: Mailed patient information — During the study year patients in this control group will receive mailed patient information about life style changes.

SUMMARY:
The hypothesis is that problem based learning (PBL) in patient education positively affects self-care agency of lifestyle changes after an event of coronary heart disease (CHD). The investigators therefore aim to determine whether long-term follow-up in primary health care in patient education involving PBL affects self-care behaviour in terms of patients' beliefs, self-efficacy and empowerment to make lifestyle changes. The general aim is to evaluate if PBL in patient education after CHD affects long-term self-care in relation to present lifestyle goals. Another aim of the study is to perform an economic assessment of long term effects of life style changes reached by using PBL after en event of CHD.

DETAILED DESCRIPTION:
Even though the convincing evidence of that self-care such as regular exercise and/or stop smoking alters the course of events after an event of coronary heart disease (CHD), risk factors remain. Outcomes can improve if core components of secondary prevention programmes are structurally pedagogically applied using adult learning principles e.g. problem based learning (PBL). Until now, most education programs for patients with CHD are not based on such principles and primary health care lacks structure in the follow-up of self-care goals of the patients. All patients will receive conventional care from their general practitioner and other care providers. They will randomly be allocated to an intervention that consists of a problem based patient education program (1 year) in PHC by trained district nurses (tutors). Patients in the control group will not attend a PBL group but receive mailed patient information during the 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages with CHD verified by MI and/or Percutaneous Coronary Intervention (PCI) and/or coronary artery by-pass surgery (CABG) within 12 months before planned start of the intervention.
* Patients should be stable regarding their cardiac conditions and have optimised cardiac medication not substantially changed during the last month, completed heart school in hospital care (if applicable), listed at one of five specific primary health care centres agreed to join the project at time of inclusion.

Exclusion Criteria:

* Planned CABG or other causes demanding continued cardiologist care; e.g. on-going contact with heart failure clinic due to drug titration or investigations e.g. myocardial scintigraphy to detect ischemia before a new PCI
* Life expectancy ≤ 1 year, documented psychiatric disease that render difficulties to cooperate with other people or obvious abuse of alcohol or narcotics.
* Patients will also be excluded if they are unable to communicate or read the Swedish language and if they participate in other studies affecting the results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
The primary-endpoint is empowerment to reach self-care goals after 5 years | At baseline and after 5 years
  Focus on empowerment to reach self-care goals will be in general, healthy food, physical activity

SECONDARY OUTCOMES:
Self-efficacy to reach self-care goals after 1 year of patient education | At baseline- and after 1, 3 and 5 years
  Self-efficacy (in general; physical exercise and healthy diet); well-being and changes in patients 'beliefs about self-care. New cardiovascular events, blood pressure, BMI, waist measurement, blood tests, costs will be calculated from a health care perspective. Resource use for conventional care and the interventions will be collected prospectively throughout the study. Questionnaires will be used to determine effectiveness (quality adjusted life years) and our goal is to perform a cost-utility analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Department of social and welfare studies, Linköping University, Norrköping, Sweden

REFERENCES:
- [Derived] Andreae C, Tingstrom P, Nilsson S, Jaarsma T, Karlsson N, Karner Kohler A. Does problem-based learning improve patient empowerment and cardiac risk factors in patients with coronary heart disease in a Swedish primary care setting? A long-term prospective, randomised, parallel single randomised trial (COR-PRIM). BMJ Open. 2023 Feb 24;13(2):e065230. doi: 10.1136/bmjopen-2022-065230. PMID 36828650
- [Derived] Kohler AK, Jaarsma T, Tingstrom P, Nilsson S. The effect of problem-based learning after coronary heart disease - a randomised study in primary health care (COR-PRIM). BMC Cardiovasc Disord. 2020 Aug 14;20(1):370. doi: 10.1186/s12872-020-01647-2. PMID 32795267
- [Derived] Karner Kohler A, Tingstrom P, Jaarsma T, Nilsson S. Patient empowerment and general self-efficacy in patients with coronary heart disease: a cross-sectional study. BMC Fam Pract. 2018 May 30;19(1):76. doi: 10.1186/s12875-018-0749-y. PMID 29843619
- [Derived] Karner A, Nilsson S, Jaarsma T, Andersson A, Wirehn AB, Wodlin P, Hjelmfors L, Tingstrom P. The effect of problem-based learning in patient education after an event of CORONARY heart disease--a randomised study in PRIMARY health care: design and methodology of the COR-PRIM study. BMC Fam Pract. 2012 Nov 20;13:110. doi: 10.1186/1471-2296-13-110. PMID 23164044